CLINICAL TRIAL: NCT03086174
Title: A Phase Ib,Open,Mono-center,Dose-escalation,Tolerability and Pharmacokinetic Study of Recombinant Humanized Anti-PD-1 mAb for Injection in Combination With Axitinib in Patients With Advanced Kidney Cancer and Melanoma
Brief Title: Tolerability and Pharmacokinetics of Toripalimab in Combination With Axitinib in Patients With Kidney Cancer and Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Junshi-JS001-008
Record Dates: First submitted 2017-03-09; First posted 2017-03-22 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Kidney Cancer Stage Iv; Advanced Melanoma
Keywords: anti-PD-1 monoclonal antibody; advanced; melanoma; kidney cancer
MeSH Terms: conditions — Kidney Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- humanized anti-PD-1monoclonal antibody (Experimental): humanized anti-PD-1 monoclonal antibody is to be injected intravenously 1mg/kg or 3mg/kg Q2w PLUS axitinib 5 mg orally Q2w until disease progresses or unacceptable tolerability occurs
  Interventions: Biological: humanized anti-PD-1 monoclonal antibody Toripalimab

INTERVENTIONS:
Biological: humanized anti-PD-1 monoclonal antibody Toripalimab — humanized anti-PD-1 monoclonal antibody Toripalimab is a programmed death-1 (PD-1) immune checkpoint inhibitor antibody, which selectively interferes with the combination of PD-1 with its ligands, PD-L1 and PD-L2, resulting in the activation of lymphocytes and elimination of malignancy theoretically.
  Other Names: JS001, TAB001

SUMMARY:
This is a phase Ib, open, mono-center, dose-escalation, tolerability and pharmacokinetic study evaluating the Recombinant Humanized Anti-PD-1 mAb for Injection in combination with Axitinib in patients with advanced kidney cancer and melanoma who have failed in routine systemic treatment.

DETAILED DESCRIPTION:
This is a phase Ib, open, mono-center, dose-escalation, tolerability and pharmacokinetic study evaluating the Recombinant Humanized Anti-PD-1 mAb for Injection in combination with Axitinib in patients with advanced kidney cancer and melanoma who have failed in routine systemic treatment.The study will be conducted in 2 parts: dose escalation and cohort expansion.

18 to 24 patients will be enrolled in dose escalation part.This part is to analyze safety and efficacy of the humanized anti-PD-1 antibody in combination with axitinib and to confirm dose-limiting toxicity (DLT), maximum tolerated dose (MTD) and recommended dose (RD). After finishing the dose escalation part, we will enroll other patients for each tumor types of recommended dose group to ensure each group have 10 patients. This part is to further analyze safety and efficacy of the humanized anti-PD-1 antibody.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female aged between 18 and 75 years are eligible;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* At least received first-line treatment but appeared disease progression or intolerance, and a diagnosis of an advanced kidney Cancer and melanoma confirmed by pathology (Remark: Treatment intolerance including 1) The main organ function of the patient is evaluated by the doctor that can not be treated by the first-line standard;2) Patients received a first-line treatment with a 3/4 adverse reaction;3) Patients reject first-line treatment, etc)
* Providing with tumor specimen (for testing the expression of PD -L1 and the infiltrating lymphocytes);
* At least 1 measurable lesion (only 1 measurable lymph node lesion is excluded) (routine CT scan >=20mm, spiral CT scan >=10mm, no prior radiation to measurable lesions)
* Predicted survival >=3 months;
* Brain or meningeal metastases must be disposed with surgery or radiation, and be stable clinically for at least 3 months (prior systemic steroids was allowed, but concurrent administration of systemic steroids with the study drug is excluded).
* Screening laboratory values must meet the following criteria（within past 14 days）:

hemoglobin ≥ 9.0 g/dL; neutrophils ≥ 1500 cells/ µL; platelets ≥ 100 x 10^3/ µL; total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; serum creatinine ≤1╳ULN，creatinine clearance >50ml/min (Cockcroft-Gault equation) INR, aPTT≤1.5 x ULN; Urine protein + 1 or less, if the urine protein > 1 +, need to collect 24 hours urinary protein determination, the total amount should be 1 gram or less

* Without systemic steroids within past 4 weeks
* Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 12 months after the last dose of study drug.
* Must have read, understood, and provided written informed consent voluntarily. Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Prior treatment with anti-PD-1/PD-L1/PD-L2 antibody and Axitinib
* Hypersensitivity to recombinant humanized anti-PD-1 monoclonal Abm or its components
* Prior antitumor therapy (including corticosteroids and immunotherapy) or participation in other clinical trials within past 4 weeks, or have not recovered from toxicities since the last treatment;
* Pregnant or nursing;
* Positive tests for HIV, HCV, HBsAg or HBcAb with positive test for HBV DNA (>500IU/ml);
* HBsAg or HBcAb with positive test for HBV DNA (>500IU/ml)
* History with active tuberculosis;
* Associated with clinical symptoms or symptomatic treatment of pleural effusion or ascites;
* Patients with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism or hypothyroidism;
* Severe, uncontrolled medical condition that would affect patients' compliance or obscure the interpretation of toxicity determination or adverse events, including active severe infection, uncontrolled diabetes, angiocardiopathy (heart failure > class II NYHA, heart block >II grade, myocardial infarction, unstable arrhythmia or unstable angina within past 6 months, cerebral infarction within past 3 months) or pulmonary disease ( interstitial pneumonia, obstructive pulmonary disease or symptomatic bronchospasm).
* Evidence with active CNS disease;
* Prior treatment with bone marrow stimulating factors，such as CSF (colony stimulating factor), EPO (erythropoietin), within past 1 weeks;
* Prior live vaccine therapy within past 4 weeks;
* Received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
* Prior major surgery within past 4 weeks (diagnostic surgery excluded).
* Psychiatric medicines abuse without withdrawal, or history of psychiatric illness.
* Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as basal cell skin cancer or carcinoma in situ of the cervix.
* Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 years
  Safety assessments including vital signs, laboratory tests, and adverse event monitoring

SECONDARY OUTCOMES:
PD-1 receptor occupancy of blood | 3 years
  To test the PD - 1 receptor share in the blood
Objective Response Rate (ORR) by irRC and RECIST 1.1 | 3 years
  The treatment effect of JS001 in combination with axitinib, will be assessed using irRC and RECIST 1.1 to determine tumor response.
Duration of Response (DOR) by irRC and RECIST 1.1 | 3 years
  The treatment effect of JS001 in combination with axitinib, will be assessed using irRC and RECIST 1.1 to determine duration of response.
Disease Control Rate (DCR) by irRC and RECIST 1.1 | 3 years
  The treatment effect of JS001 in combination with axitinib, will be assessed using irRC and RECIST 1.1 to determine disease control rate.
Time to response (TTR) by irRC and RECIST 1.1 | 3 years
  The treatment effect of JS001 in combination with axitinib, will be assessed using irRC and RECIST 1.1 to determine time to response.
Progression-free survival(PFS) by irRC and RECIST 1.1 | 3 years
  The treatment effect of JS001 in combination with axitinib, will be assessed using irRC and RECIST 1.1 to determine progression-free survival time.
Overall survival (OS) by irRC and RECIST 1.1 | 3 years
  The treatment effect of JS001 in combination with axitinib, will be assessed using irRC and RECIST 1.1 to determine overall survival.
PK Parameter: Maximum Plasma Concentration (Cmax) | 3 years
  Maximum Plasma Concentration (Cmax) after single dose injection of Anti-PD-1 Monoclonal Antibody (mAb) in combination with axitinib
PK Parameter: Peak Time (Tmax) | 3 years
  Peak Time (Tmax) after single dose injection of Anti-PD-1 mAb in combination with axitinib
PK Parameter: t1/2 | 3 years
  t1/2 after single dose injection of Recombinant Humanized Anti-PD-1 mAb in combination with axitinib
PK Parameter: Area Under the Curve (AUC) | 3 years
  Area Under the Curve (AUC) after single dose injection of Anti-PD-1 mAb in combination with axitinib
PK Parameter: Plasma clearance (CL) | 3 years
  Plasma clearance (CL) after single dose injection of Anti-PD-1 mAb in combination with axitinib
PK Parameter: Apparent volume of distribution (V) | 3 years
  Apparent volume of distribution (V) after single dose injection of Anti-PD-1 mAb in combination with axitinib
PK Parameter: Minimum Plasma Concentration (Cmin) | 3 years
  Minimum Plasma Concentration (Cmin) of steady state after multiple dose injection of Anti-PD-1 mAb in combination with axitinib
PK Parameter: Average Plasma Concentration (Cav) | 3 years
  Average Plasma Concentration (Cav) of steady state after multiple dose injection of Anti-PD-1 mAb in combination with axitinib
PK Parameter: degree of fluctuation (DF) | 3 years
  degree of fluctuation (DF) of steady state after multiple dose injection of Anti-PD-1 mAb in combination with axitinib
PK Parameter: Apparent volume of distribution of steady state (Vss) | 3 years
  Apparent volume of distribution of steady state (Vss) after multiple dose injection of Anti-PD-1 mAb in combination with axitinib

OTHER OUTCOMES:
correlation analysis of PD-L1 expression of tumor and ORR | 3 years
  correlation analysis of PD-L1 expression of tumor and objective response rate
correlation analysis of PD-L1 expression of tumor and DOR | 3 years
  correlation analysis of PD-L1 expression of tumor and duration of response
correlation analysis of PD-L1 expression of tumor and DCR | 3 years
  correlation analysis of PD-L1 expression of tumor and disease control rate
correlation analysis of PD-L1 expression of tumor and TTR | 3 years
  correlation analysis of PD-L1 expression of tumor and time to response
correlation analysis of PD-L1 expression of tumor and PFS | 3 years
  correlation analysis of PD-L1 expression of tumor and progression-free survival
correlation analysis of PD-L1 expression of tumor and OS | 3 years
  correlation analysis of PD-L1 expression of tumor and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Rini BI, Escudier B, Tomczak P, Kaprin A, Szczylik C, Hutson TE, Michaelson MD, Gorbunova VA, Gore ME, Rusakov IG, Negrier S, Ou YC, Castellano D, Lim HY, Uemura H, Tarazi J, Cella D, Chen C, Rosbrook B, Kim S, Motzer RJ. Comparative effectiveness of axitinib versus sorafenib in advanced renal cell carcinoma (AXIS): a randomised phase 3 trial. Lancet. 2011 Dec 3;378(9807):1931-9. doi: 10.1016/S0140-6736(11)61613-9. Epub 2011 Nov 4. PMID 22056247
- [Background] Du Four S, Maenhout SK, De Pierre K, Renmans D, Niclou SP, Thielemans K, Neyns B, Aerts JL. Axitinib increases the infiltration of immune cells and reduces the suppressive capacity of monocytic MDSCs in an intracranial mouse melanoma model. Oncoimmunology. 2015 Jan 22;4(4):e998107. doi: 10.1080/2162402X.2014.998107. eCollection 2015 Apr. PMID 26137411
- [Derived] Li S, Wu X, Yan X, Zhou L, Chi Z, Si L, Cui C, Tang B, Mao L, Lian B, Wang X, Bai X, Dai J, Kong Y, Tang X, Feng H, Yao S, Flaherty KT, Guo J, Sheng X. Toripalimab plus axitinib in patients with metastatic mucosal melanoma: 3-year survival update and biomarker analysis. J Immunother Cancer. 2022 Feb;10(2):e004036. doi: 10.1136/jitc-2021-004036. PMID 35193932